CLINICAL TRIAL: NCT00175656
Title: Titanium Elastic Nails in the Treatment of Paediatric Femoral Fractures: A Prospective Randomized Clinical Trial of Eliminating Nail Protrusion to Decrease Soft Tissue Complications
Brief Title: Titanium Elastic Nails in the Treatment of Pediatric Femur Fractures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Christopher Reilly, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H03-70522; W03-0165
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Femur Fracture
Keywords: Femur fracture; titanium elastic nails
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Elimination of titanium elastic nail prominence at the insertion site and leaving the nails in situ — See Detailed Description.

SUMMARY:
Titanium elastic nails in the pediatric femoral fractures: A prospective randomized clinical trial of eliminating nail protrusion to decrease soft tissue complications

DETAILED DESCRIPTION:
This study will be conducted as a prospective cohort study of children and adolescents treated with TEN for a femoral shaft fracture. All children and adolescents presenting to the Emergency department of a participating center with a femur fracture will be approached for inclusion in the study. The primary outcome for this study will be functional recovery, as measured using a pediatric specific generic QOL measurement tool. The clinical outcome measure which will be used will be the performance version of the ASK (ASK-p) which has been previously tested and shown to be valid, reliable, and responsive in children and adolescents with acute and chronic Orthopaedic disorders. The first time point for data collection will be at four months. Clinical data which will be obtained over the course of follow-up will include clinical evaluation of hip and knee range of motion, limb rotation, clinical measurement of limb length, fracture union, and the presence of complications, including the need for nail removal in the group in which it was not planned. The second time point for data collection will be at one year. Again, the ASK-p will be mailed to all subjects in advance to allow completion at the desired time. The return of questionnaires and process for reminder notifications will proceed in a similar fashion to the four month time point. Clinical and radiographic data will be collected in a similar fashion to the four month time point. No subjects will be excluded on the basis of failure to return questionnaires at the one year time point since this represents a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

open femoral physes; closed midshaft femur fracture; no concomitant injuries to either lower extremity; no history of injury to either femur; no history of asymmetric femoral malalignment; agree to participate in 2 years of follow up; informed consent/assent.

Exclusion Criteria:

open midshaft femur fractures; other injuries to either lower extremity; a history of injury to either femur; unable to comply with 2 years of follow-up

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To investigate the soft tissue complication rate and to determine the clinical and functional outcomes at 4 months following femoral fracture reduction using titanium elastic nails in skeletally immature patients. | 4 months

SECONDARY OUTCOMES:
To compare the clinical and functional outcomes between leaving the nails in situ and removing them; 1 year and 2 year follow-up. | 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Reilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada